CLINICAL TRIAL: NCT02061332
Title: A Randomized Trial of HER-2/Neu Pulsed DC1 Vaccine for Patients With DCIS
Brief Title: DC Vaccine for Patients With Ductal Carcinoma In Situ
Acronym: DCIS6
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 807010; 15107 (Other: CTSRMC, Abramson Cancer Center, University of Pennsylvania); NCT00923143 (obsolete NCT alias)
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer; DCIS
Keywords: Breast Cancer; DCIS; Immunotherapy; Vaccine; Dendritic Cell
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intranodal Vaccine (Experimental): An ultrasound device (probe) will be placed over the area of the groin or armpit. The vaccine needle will then be placed under the probe, and guided by the ultrasound machine to the groin lymph nodes or axillary nodes. You will be given a HER-2 pulsed dendritic cell vaccine in two different groin lymph nodes or axillary nodes per visit. Each dose will consist of 1.0-2.0 x 107 cells and will be injected into 1-2 different groin lymph nodes or axillary nodes.
  Interventions: Biological: HER-2 Pulsed Dendritic cell Vaccine
- Intralesional Vaccine (Experimental): The HER-2 pulsed dendritic cell vaccine will be directly injected into the quadrant of the breast affected with DCIS. The location will be determined by referring to the patient's mammogram. Each dose will consist of 1.0-2.0 x 107 cells and will be injected into the quadrant of the breast affected with DCIS.
  Interventions: Biological: HER-2 Pulsed Dendritic cell Vaccine
- Intranodal + Intralesional Vaccine (Experimental): You will be given a HER-2 pulsed dendritic cell vaccine in two different groin lymph nodes or axillary nodes and the quadrant of the breast affected with DCIS. An ultrasound device (probe) will be placed over the groin or armpit. The vaccine needle will be placed under the probe, and guided by the ultrasound machine to the groin lymph nodes or axillary nodes. The intralesional vaccine will be directly injected into the quadrant of the breast affected with DCIS. The location will be determined by referring to the patient's mammogram. Each dose will consist of 1.0-2.0 x 107 cells. Approximately half of the dose will be injected into 1-2 different groin lymph nodes or axillary nodes. The remaining half will be injected into the quadrant of the breast affected with DCIS.
  Interventions: Biological: HER-2 Pulsed Dendritic cell Vaccine

INTERVENTIONS:
Biological: HER-2 Pulsed Dendritic cell Vaccine — 6 weekly HER-2 pulsed dendritic cell vaccines will be administered to subjects in each of the 3 arms.

SUMMARY:
Women who are diagnosed with Her-2/neu over-expressing DCIS will receive DC1 vaccines by intranodal, intralesional, or both routes of administration. The primary objective will be safety and administration with secondary objectives of immune activation and clinical response.

DETAILED DESCRIPTION:
The treatment of patients with DCIS can be individualized and tailored to the type of DCIS and the relative risk of the lesion. HER-2/neu over-expressing DCIS represents a group of patients with significant risk for development of invasive breast cancer. In this proposal we will continue to evaluate the development of type I polarized DC for the treatment of DCIS by evaluating whether further improvements in therapeutic response can be achieved by intratumoral administration of HER-2/neu pulsed DC1 compared with our current intranodal administration. Women who are diagnosed with Her-2/neu over-expressing DCIS with no invasive carcinoma will be eligible for this study. Patients will receive DC1 vaccines by intranodal, intralesional, or both routes of administration. The primary objective will be safety and administration with secondary objectives of immune activation and clinical response. We will also develop a novel assay to monitor ongoing immunity to HER-2/neu, and lastly will begin to develop these vaccines for patients with invasive breast cancer as well. Fifty-four subjects will be randomized to one of three treatment arms: intranodal injection, intralesional injection, or intranodal and intralesional injection of the vaccine. Upon entering this study, the subjects' blood will be drawn in a way that collects only the white blood cells. Subjects then receive six vaccines over a six week period. They will then undergo the standard surgical procedure to remove any remaining DCIS in the breast.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Subjects with biopsy-proven DCIS, DCIS with microinvasion, DCIS with invasive disease under 5 mm, or Paget's Disease of the nipple (DCIS of the nipple) who have not yet received definitive treatment.
* HER-2/neu positive tumor as determined by >5% of tumor population expressing this marker by immunohistochemical staining 2+ using anti-HER-2/neu verified by Dr. Paul Zhang in the Department of Pathology.
* Women of childbearing age with a negative pregnancy test documented prior to enrollment.
* Subjects with ECOG Performance Status Score of 0 or 1 (Appendix D).
* Subjects willing to use birth control if necessary
* Subjects who have voluntarily signed a written Informed Consent in accordance with institutional policies after its contents have been fully explained to them.

Exclusion Criteria:

* Pregnant or lactating females (pregnancy testing to be performed within 7 days prior to administration of first dose of vaccine).
* Subjects who have had a complete excisional biopsy of their tumor.
* Subjects with suspicion of invasive disease > 5mm by MRI performed within 2 months of study recruitment.
* Screen and exclude subjects with positive HIV or hepatitis C at baseline.
* Subjects with coagulopathies, including thrombocytopenia with platelet count <75,000, INR > 1.5 and partial thromboplastin time > 50 sec
* Subjects with major cardiac illness MUGA < 50% EF.
* Subjects with pre-existing medical illnesses or medications which might interfere with the study.
* Subjects with laboratory tests reflecting ¬> grade 1 toxicity by NCI CTC version 3.0 including CBC, liver function tests, urinalysis, EKG if cannot be corrected on repeat test in 7 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2014-08-08 (Actual); Study Completion 2015-10-07 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | up to 60 minutes post vaccine
  Blood pressure will be obtained just prior to the vaccination then, every 15 minutes for the first hour after the dose is given.
Temperature | up to 60 minutes post vaccine
  Temperature will be obtained just prior to the vaccination then, every 15 minutes for the first hour after the dose is given.
Pulse | up to 60 minutes post vaccine
  Pulse will be obtained just prior to the vaccination then, every 15 minutes for the first hour after the dose is given.

SECONDARY OUTCOMES:
Immune Response | 6-8 weeks
  Subjects will undergo leukapheresis after completion of 6 vaccines and 3 boost vaccines for the purpose of obtaining lymphocytes and monocytes for in vitro immunologic testing.
Mammogram | 6-8 weeks
  All subjects will have a post-vaccine bilateral mammogram to evaluate response to vaccination. Mammograms will be performed within two weeks after the 6th vaccination.
MRI | 6-8 weeks
  All subjects will have a post-vaccine bilateral breast MRI to evaluate response to vaccination. MRIs will be performed within two weeks after the 6th vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Czerniecki, M.D., Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Czerniecki BJ, Roses RE, Koski GK. Development of vaccines for high-risk ductal carcinoma in situ of the breast. Cancer Res. 2007 Jul 15;67(14):6531-4. doi: 10.1158/0008-5472.CAN-07-0878. PMID 17638860
- [Background] Czerniecki BJ, Koski GK, Koldovsky U, Xu S, Cohen PA, Mick R, Nisenbaum H, Pasha T, Xu M, Fox KR, Weinstein S, Orel SG, Vonderheide R, Coukos G, DeMichele A, Araujo L, Spitz FR, Rosen M, Levine BL, June C, Zhang PJ. Targeting HER-2/neu in early breast cancer development using dendritic cells with staged interleukin-12 burst secretion. Cancer Res. 2007 Feb 15;67(4):1842-52. doi: 10.1158/0008-5472.CAN-06-4038. Epub 2007 Feb 9. PMID 17293384
- [Background] Koski GK, Koldovsky U, Xu S, Mick R, Sharma A, Fitzpatrick E, Weinstein S, Nisenbaum H, Levine BL, Fox K, Zhang P, Czerniecki BJ. A novel dendritic cell-based immunization approach for the induction of durable Th1-polarized anti-HER-2/neu responses in women with early breast cancer. J Immunother. 2012 Jan;35(1):54-65. doi: 10.1097/CJI.0b013e318235f512. PMID 22130160
- [Background] Sharma A, Koldovsky U, Xu S, Mick R, Roses R, Fitzpatrick E, Weinstein S, Nisenbaum H, Levine BL, Fox K, Zhang P, Koski G, Czerniecki BJ. HER-2 pulsed dendritic cell vaccine can eliminate HER-2 expression and impact ductal carcinoma in situ. Cancer. 2012 Sep 1;118(17):4354-62. doi: 10.1002/cncr.26734. Epub 2012 Jan 17. PMID 22252842